CLINICAL TRIAL: NCT05250921
Title: The Effect of Corticision on Perceived Pain and Discomfort for Patients With Crowded Lower Anterior Teeth in Young Adult Patients: Randomized Clinical Trial
Brief Title: Evaluation of the Patient Experience With a Surgically-assisted Acceleration Method of Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-03-2022
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Crowding, Tooth
Keywords: Corticision; Visual analog scale; Mild and moderate crowding; Surgical blade; Pain; Discomfort
MeSH Terms: conditions — Malocclusion; Lymphoma, Follicular; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticision (Experimental): Corticision will be performed on the lower anterior teeth using a surgical blade and a hammer.
  Interventions: Procedure: Corticision
- Conventional method (Active Comparator): A fixed appliance will be applied using conventional braces without any surgical procedure.
  Interventions: Device: Conventional fixed appliance

INTERVENTIONS:
Procedure: Corticision — Corticision will be performed to enhance teeth alignment.
  Arms: Corticision
Device: Conventional fixed appliance — No surgical intervention is going to be applied to the patients in this group.
  Arms: Conventional method

SUMMARY:
The duration of orthodontic treatment is one of the exacerbation causes of orthodontic pain. Several methods have been suggested to reduce the duration of orthodontic treatment classified to surgical and non-surgical methods.

Researches used minimally invasive surgical methods like corticision, piezocesion, disicion, micro-osteoperforation, and piezopuncture indicated that most of these methods can accelerate dental movement by 20 - 40% without causing additional pain as a result of using those methods.

Applying corticision on the lower anterior teeth using a surgical blade and a hammer may accelerate tooth alignment during orthodontic treatment. This study consists of two groups, patients will be randomly assigned to one of these two groups.

DETAILED DESCRIPTION:
Pain is defined as an unpleasant emotional sensory experience associated with actual or potential harm. It was mentioned as one of the most common complaints related to orthodontic treatment, and around 65-95% of patients undergoing orthodontic treatment suffer from various degrees of pain.

Corticision is one of the minimally invasive surgical procedures that is not associated with flap lifting. It was used to accelerate tooth movement in animals and case report studies. Its application on humans may aggravate their fear and anxiety towards the pain that may accompany this technique.

No study in the literature has been searched in patient perception of pain, discomfort, levels of acceptance and satisfaction accompanied corticision application application, but in this study, these previous variables accompanied corticision technique have been studied on crowded lower anterior teeth cases which are one of the most common types of malocclusions.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 18 and 24 years
2. Completion of permanent dentition (except third molars)
3. Mild to moderate crowding (2-6 mm according to Little's index)
4. Absence of medications intake that interferes with pain perception for at least one week before the beginning of the treatment

Exclusion Criteria:

1. Systematic diseases that could affect bone and tooth movement and no contraindication avoid oral surgery
2. Medical conditions that affect tooth movement (Corticosteroid, NSAIDs)
3. Patients had previous orthodontic treatments
4. Poor oral hygiene or concurrent periodontal disease

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Change in the levels of pain | at 1, 7, 14 days following the onset of orthodontic treatment
  Pain is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of pain being experienced. The left end of the line refers to no pain (VAS=0) where the right end refers to maximum (unimaginable) pain (VAS=100). The level of pain is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the pain.
Change in the levels of discomfort: | at 1, 7, 14 days following the onset of orthodontic treatment
  discomfort is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of discomfort being experienced. The left end of the line refers to no discomfort (VAS=0) where the right end refers to maximum discomfort (VAS=100). The level of discomfort is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the discomfort.
Change in the levels of swelling | at 1, 7, 14 days following the onset of orthodontic treatment
  swelling is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of swelling being experienced. The left end of the line refers to no swelling (VAS=0) where the right end refers to maximum swelling (VAS=100). The level of swelling is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the swelling.
Change in the perception of mastication problems: | at 1, 7, 14 days following the onset of orthodontic treatment
  difficulties of mastication are assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of difficulties in mastication being experienced. The left end of the line refers to no difficulties (VAS=0) where the right end refers to maximum difficulties (VAS=100). The level of difficulties in mastication are represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the difficulties of mastication.
Number of analgesic tables taken | at seven days following the onset of orthodontic treatment
  The number of tablets used: Patients in both groups were asked about taking analgesics and their quantity (mg) They answered about taking analgesics using a two-point scale (1. Yes or 2. No), and their quantity by mentioning how many tablets they took.

SECONDARY OUTCOMES:
Satisfaction using VAS: | At the end of leveling and alignment
  Definition: satisfaction is assessed for both groups by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of satisfaction. The left end of the line refers to no satisfaction (VAS=0) where the right end refers to maximum satisfaction (VAS=100). The level of satisfaction is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the satisfaction.
Satisfaction with the ease of the procedure | At the end of leveling and alignment
  is assessed for both groups by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of ease. The left end of the line refers to no ease (VAS=0) where the right end refers to maximum ease (VAS=100). The grade of ease is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the ease of the procedure.
Satisfaction through acceptability of the procedure | At the end of leveling and alignment
  Patients in corticision group were asked about possibility of repeating the procedure, and they answered using a two-point scale (1. Yes or 2. No).
Satisfaction through recommending the procedure | At the end of leveling and alignment
  Recommendation to a friend: Patients in corticision group were asked about making recommendation to a friend, and they answered using a two-point scale (1. Yes or 2. No).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Radwan Sirri, DDS MSc, Principal Investigator — Department of orthodontics, Damascus University, Syria; Ahmad S Burhan, DDS MSc PhD, Study Director — Professor of Orthodontics, Department of Orthodontics, University of Damascus Dental School; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Professor of Orthodontics, Department of Orthodontics, University of Damascus Dental School; Fehmieh R Nawaya, DDS MSc PhD, Study Director — Associate Professor, Department of Pediatric Dentistry,Syrian PrivateUniversity; Rashad MT Murad, DDS MSc PhD, Study Director — Professor of Toxins and Pharmaceutics, University of Damascus, Faculty of Pharmacology
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984
- [Background] Alkebsi A, Al-Maaitah E, Al-Shorman H, Abu Alhaija E. Three-dimensional assessment of the effect of micro-osteoperforations on the rate of tooth movement during canine retraction in adults with Class II malocclusion: A randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2018 Jun;153(6):771-785. doi: 10.1016/j.ajodo.2017.11.026. PMID 29853235
- [Background] Charavet C, Lecloux G, Bruwier A, Rompen E, Maes N, Limme M, Lambert F. Localized Piezoelectric Alveolar Decortication for Orthodontic Treatment in Adults: A Randomized Controlled Trial. J Dent Res. 2016 Aug;95(9):1003-9. doi: 10.1177/0022034516645066. Epub 2016 Apr 29. PMID 27129491
- [Background] Yavuz MC, Sunar O, Buyuk SK, Kantarci A. Comparison of piezocision and discision methods in orthodontic treatment. Prog Orthod. 2018 Oct 29;19(1):44. doi: 10.1186/s40510-018-0244-y. PMID 30370430
- [Background] Uribe F, Davoody L, Mehr R, Jayaratne YSN, Almas K, Sobue T, Allareddy V, Nanda R. Efficiency of piezotome-corticision assisted orthodontics in alleviating mandibular anterior crowding-a randomized clinical trial. Eur J Orthod. 2017 Nov 30;39(6):595-600. doi: 10.1093/ejo/cjw091. PMID 28371882